CLINICAL TRIAL: NCT00222365
Title: Homeopathy Assessment in Terms of the Consumption of Analgesics After Knee Ligamentoplasty
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCIC 03 10
Record Dates: First submitted 2005-09-14; First posted 2005-09-22 (Estimated); Last update posted 2006-11-14 (Estimated); Status verified 2006-07

CONDITIONS: Pain
Keywords: homeopathy; assessment; pain; ligamentoplasty
MeSH Terms: conditions — Pain | interventions — Arnicae flos extract; Hypericum extract LI 160

INTERVENTIONS:
Drug: Arnica montana, 5 CH
Drug: Bryonia alba, 5 CH
Drug: Hypericum perforatum, 5 CH
Drug: Ruta graveolens, 3 DH

SUMMARY:
This is an add-on, double blind, and randomised clinical trial with three groups: a homeopathic group, a placebo group, and a temporal control group.

The aim of this trial is to assess the effect of homeopathy on the consumption of morphine delivered by PCA (patient control analgesia) for 24 hours after a knee ligamentoplasty.

DETAILED DESCRIPTION:
We test the effectiveness of an homeopathic drug versus placebo and a temporal control group (patient with no add-on treatment) following orthopedic knee surgery.

All patients have a PCA of morphine for 24 hours after surgery. After this period they can take an oral tablet of morphine on request.

Group A: Patients with study treatment (homeopathy) allocation. Double blind group with 70 patients

Group B: Patients with placebo allocation. Double blind group with 70 patients

Group C: Temporal control group with patients who take only the morphine. Open group with 25 patients

The total power: 70 +70 + 25 = 165 patients

Main Objective:

* To assess the effect of homeopathy in terms of morphine consumption delivered by PCA (patient control analgesia) for 24 hours after a knee ligamentoplasty.

Secondary Objectives:

* To assess the effect of homeopathy in terms of total morphine consumption between H24 and H72 after a knee ligamentoplasty.
* To assess the effect of homeopathy on the pain perception using a analogical visual scale for 72 hours.
* To asses the placebo effect of the homeopathic treatment.

Main Assessment Criterion:

* Morphine consumption delivered by PCA between 0 and 24 hours after knee ligamentoplasty

Secondary Assessment Criteria:

* Morphine consumption between 0 and 72 hours after ligamentoplasty
* Pain assessment at H0, H4, H24 and H72 using 10 cm Analogical Visual Scale

Inclusion Criteria:

* age ranging from 18 to 60.
* patients candidates for a ligamentoplasty of the anterior cruciate ligament.

Exclusion Criteria:

* patient with corticoid and immunodepressor treatment

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 18 to 60 years.
* Patients who are candidates for a ligamentoplasty of the anterior cruciate ligament.

Exclusion Criteria:

* Patients with corticoid and immunodepressor treatment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165
Dates: Start 2003-12; Study Completion 2006-05

PRIMARY OUTCOMES:
Morphine consumption delivered by PCA between 0 and 24 hours after a knee ligamentoplasty

SECONDARY OUTCOMES:
Morphine consumption between 0 and 72 hours after the ligamentoplasty
Pain assessment at hour 0 (H0), H4, H24 and H72 with 10 cm Analogical Visual Scale

CONTACTS AND LOCATIONS:
Overall Officials: CRACOWSKI Jean-Luc, Dr, Principal Investigator — Clinical Trial Center
Locations (1):
- University Hospital of Grenoble, Grenoble, France

REFERENCES:
- [Background] Barnes J, Resch KL, Ernst E. Homeopathy for postoperative ileus? A meta-analysis. J Clin Gastroenterol. 1997 Dec;25(4):628-33. doi: 10.1097/00004836-199712000-00016. PMID 9451677
- [Background] Ernst E. A systematic review of systematic reviews of homeopathy. Br J Clin Pharmacol. 2002 Dec;54(6):577-82. doi: 10.1046/j.1365-2125.2002.01699.x. PMID 12492603
- [Background] Linde K, Clausius N, Ramirez G, Melchart D, Eitel F, Hedges LV, Jonas WB. Are the clinical effects of homeopathy placebo effects? A meta-analysis of placebo-controlled trials. Lancet. 1997 Sep 20;350(9081):834-43. doi: 10.1016/s0140-6736(97)02293-9. PMID 9310601
- [Background] Lokken P, Straumsheim PA, Tveiten D, Skjelbred P, Borchgrevink CF. Effect of homoeopathy on pain and other events after acute trauma: placebo controlled trial with bilateral oral surgery. BMJ. 1995 Jun 3;310(6992):1439-42. doi: 10.1136/bmj.310.6992.1439. PMID 7613277
- [Result] Cucherat M, Haugh MC, Gooch M, Boissel JP. Evidence of clinical efficacy of homeopathy. A meta-analysis of clinical trials. HMRAG. Homeopathic Medicines Research Advisory Group. Eur J Clin Pharmacol. 2000 Apr;56(1):27-33. doi: 10.1007/s002280050716. PMID 10853874